CLINICAL TRIAL: NCT04602689
Title: Effectiveness of Fibrin Glue to Prevent Bleeding in High-risk Patients After Endoscopic Submucosal Dissection in Gastric Neoplasm : A Prospective Randomized Controlled Study
Brief Title: Fibrin Glue After ESD for High Risk Patients of Bleeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Soo-Jeong Cho, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2004-093-1117
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Early Gastric Cancer; Gastric Adenoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fibrin glue group (Experimental): Spread Fibrin glue(Greenplast Q™) at iatrogenic ulcer after gastric ESD
  Interventions: Drug: Human fibrinogen concentrate
- Control group (No Intervention): No intervention after gastric ESD

INTERVENTIONS:
Drug: Human fibrinogen concentrate — Spread the Human fibrinogen concentrate/Aprotinin/Thrombin/Calcium chloride hydrate mixture on iatrogenic ulcer after ESD
  Arms: Fibrin glue group

SUMMARY:
It is a prospective randomized controlled study to look for effectiveness of fibrin glue to prevent bleeding in high-risk patients after endoscopic submucosal dissection in gastric neoplasm.

DETAILED DESCRIPTION:
Investigators want to observe the bleeding rate after endoscopic submucosal dissection for gastric tumors in the high-risk group of bleeding (the size of the iatrogenic ulcer is expected to be 40mm or more, or taking aspirin, antiplatelet drugs, and anticoagulants).

After resection and hemostasis with ESD, Fibrin glue (Greenplast Q™) is applied to the iatrogenic ulcer at the end of the procedure, and the control group will not be applied.

After that, observe whether there is a difference in the bleeding rate within 48 hours and 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-1
* Patients scheduled to undergo ESD due to gastric tumor (dysplasia, early gastric cancer)
* Patients who are expected to have an iatrogenic ulcer size of 40mm or more after endoscopic submucosal dissection, or are taking aspirin, antiplatelet drugs, or anticoagulants
* Patients who show adequate patient compliance and have adequate geographic distance for follow-up observation.

Exclusion Criteria:

* Patients with sensitivity to cow protein or its derived ingredients
* Patients who had previously undergone partial gastrectomy
* Patients with early gastric cancer at the site previously undergoing ESD
* Patients with clinically significant cardiopulmonary disease
* Patients with active hepatitis, liver disease that is not well controlled by treatment, or severe liver disorder
* Patients with severe renal impairment
* Patients with severe bone marrow dysfunction
* Patients with severe blood clotting impairment (including hemophilia)
* Patients with serious neurological or mental illness (e.g. epilepsy or dementia)
* Patients with reported side effects of contrast media
* Pregnant and lactating women
* Patients who have not obtained the informed consent of the patient and guardian
* Patients who are inadequate for clinical trials as judged by the attending physician

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Bleeding after ESD | 4 weeks
  Number of gastrointestinal bleeding events within 4 weeks after the procedure

SECONDARY OUTCOMES:
Early bleeding after ESD | 48 hours
  Number of gastrointestinal bleeding events within 48 hours after the procedure
Delayed bleeding after ESD | from 48 hours to 4 weeks
  Number of gastrointestinal bleeding events from 48 hours to 4 weeks after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eunwoo Lee, M.D., Study Director — fellowship
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee HD, Lee E, Kim SG, Shin CM, Park JC, Choi KD, Hahn S, Cho SJ. A Randomized Controlled Trial of Fibrin Glue to Prevent Bleeding After Gastric Endoscopic Submucosal Dissection. Am J Gastroenterol. 2023 May 1;118(5):892-899. doi: 10.14309/ajg.0000000000002172. Epub 2022 Dec 30. PMID 36594814